CLINICAL TRIAL: NCT00569400
Title: Comparison of Efficacy and Safety of Human Insulin Produced by the Current Process and the NN729 Process in Type 1 Diabetes Mellitus
Brief Title: Comparison of Human Insulin Produced by the Current Process and the NN729 Process in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN729-1541
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: human insulin

SUMMARY:
This trial is conducted in Asia and Oceania. The aim of this trial is to compare the efficacy and safety of human insulin produced by the current process and the NN729 process in type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Duration of diabetes for at least 12 months
* Basal/bolus treatment with human insulin for at least 2 months preceding trial start
* Body Mass Index (BMI) lesser than or equal to 35.0 kg/m2
* HbA1c lesser than or equal to 12.0%

Exclusion Criteria:

* Proliferative retinopathy or maculopathy requiring acute treatment or laser treatment within the last 6 months
* Any condition that the investigator and/or sponsor feel would interfere with trial participation
* Known or suspected allergy against trial product or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2003-05-01 (Actual); Primary Completion 2004-01-19 (Actual); Study Completion 2004-01-19 (Actual)

PRIMARY OUTCOMES:
Change of human insulin antibodies | after 26 weeks of treatment

SECONDARY OUTCOMES:
Change of human insulin antibodies
Frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (15):
- Australia (7):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, Dunedin
  - Novo Nordisk Investigational Site, Hamilton
  - Novo Nordisk Investigational Site, Kippa-Ring
  - Novo Nordisk Investigational Site, Miranda
  - Novo Nordisk Investigational Site, Stones Corner
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Malaysia (3):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Georgetown, Penang
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
- Philippines (4):
  - Novo Nordisk Investigational Site, Cebu City
  - Novo Nordisk Investigational Site, Iloilo City
  - Novo Nordisk Investigational Site, Makati City
  - Novo Nordisk Investigational Site, Marikina City

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com